CLINICAL TRIAL: NCT04207775
Title: Real World Molecular Testing, Treatment Patterns, and Clinical Outcomes in EGFR Mutation-Positive, Locally Advanced or Metastatic Chinese NSCLC Patients, Who Have Progressed From First-line EGFR-TKI Therapy (PISCES)
Brief Title: Real World Study in Locally Advanced or Metastatic NSCLC Patients, Progressed From First-line EGFR-TKI Therapy
Acronym: PISCES
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D5160R00031
Record Dates: First submitted 2019-12-19; First posted 2019-12-23 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Locally Advanced or Metastatic NSCLC
Keywords: NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- NSCLC: Patients with confirmed EGFR mutation-positive, locally advanced or metastatic NSCLC, who have progressed from first line EGFR-TKI therapy who will receive different treatment

SUMMARY:
To estimate parameters associated with treatment patterns and related clinical outcomes.Including physician reported PFS and OS.

DETAILED DESCRIPTION:
The objectives of this study are to assess molecular testing, treatment patterns, and associated clinical outcomes among patients with epidermal growth factor receptor (EGFR) mutation-positive locally advanced or metastatic non-small cell lung cancer (NSCLC) who have progressed from first-line EGFR-TKI (tyrosine kinase inhibitor) therapy. This study is descriptive in nature and does not attempt to test any specific a priori hypotheses

ELIGIBILITY:
Inclusion Criteria

1. Male or female patients with age ≥18 years old
2. Histologically or cytologically confirmed locally advanced or metastatic NSCLC patients
3. Patients with prior confirmed EGFR mutation-positive, who have progressed from first line EGFR-TKI*
4. Provision of written informed consent by the patient should be within 6 weeks of the date of progression from first line EGFR-TKI treatment *Note：

   1. First-line EGFR-TKI is monotherapy;
   2. EGFR-TKI has been launched in China includes first-generation, second-generation or third-generation EGFR-TKI, but not including the original chemical compound
   3. Exclude the Chinese traditional medicine that is being used to treat lung cancer
   4. Progression was determined according to Recist1.1 criteria.

Exclusion Criteria

1. Involvement in the planning and/or conduct of the other intervention study
2. Previous enrolment in the present study
3. Pregnancy or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult male or female patients (with age ≥18 years old) who have given provision of signed and dated written informed consent by the patient or legally acceptable Patients with confirmed EGFR mutation-positive, locally advanced or metastatic NSCLC, who have progressed from first line EGFR-TKI therapy
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2020-03-30 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Physician-reported clinical outcomes, PFS | From enrolment to follow-up of up to 36 months
  from date of second-line treatment initiation until progression by RECIST1.1 criteria, or death
Physician-reported clinical outcomes, OS | From enrolment to follow-up of up to 36 months
  the date of second-line treatment initiation until death from any cause(only for patients receiving 2L CT and 2L TKI, separately)
Time to initiate second line therapy from progression from 1L treatment | From enrolment to follow-up of up to 36 months
  Time to initiate second line therapy from RECIST1.1 defined progression from 1L treatment
Response rate | From enrolment to follow-up of up to 36 months
  Response rate reported by physician or judged by Recist1.1 after receiving any pattern of therapy
chemotherapy | From enrolment to follow-up of up to 36 months
  For each line of chemotherapy received but not limited in:Therapy regimen，Therapy duration measured as time from therapy start date to time of therapy end date，Number of cycles received，Reason for cessation of therapy
immunotherapy | From enrolment to follow-up of up to 36 months
  For each line of immunotherapy received but not limited in:Therapy regimen，Therapy duration measured as time from therapy start date to time of therapy end date，Number of cycles received，Reason for cessation of therapy
targeted therapy | From enrolment to follow-up of up to 36 months
  For each line of targeted therapy received but not limited in:Therapy regimen，Therapy duration measured as time from therapy start date to time of therapy end date，Number of cycles received，Reason for cessation of therapy
local therapy | From enrolment to follow-up of up to 36 months
  For each line of local therapy received but not limited in:Therapy regimen，Therapy duration measured as time from therapy start date to time of therapy end date，Number of cycles received，Reason for cessation of therapy
palliative/supportive care | From enrolment to follow-up of up to 36 months
  Any palliative/supportive care received

SECONDARY OUTCOMES:
Molecular testing sample type | From enrolment to follow-up of up to 36 months
  To estimate parameters in the target population associated with molecular testing patterns, including molecular testing sample type
Molecular test outcome | From enrolment to follow-up of up to 36 months
  To estimate parameters in the target population associated with molecular testing patterns, including molecular test outcome
changes in testing rate over time | From enrolment to follow-up of up to 36 months
  To estimate parameters associated with molecular testing patterns, including changes in testing rate over time
Molecular testing rate | From enrolment to follow-up of up to 36 months
  Molecular testing rate defined as the number of patients identified as having received molecular testing divided by the number of patients
Time from progression date to molecular testing | From enrolment to follow-up of up to 36 months
  Time from the RECIST defined progression date to molecular testing
Molecular testing method of biopsy | From enrolment to follow-up of up to 36 months
  To estimate parameters in the target population associated with molecular testing patterns, including molecular testing method of biopsy
Molecular testing turnaround time | From enrolment to follow-up of up to 36 months
  To estimate parameters in the target population associated with molecular testing patterns, including molecular testing turnaround time
Molecular test type | From enrolment to follow-up of up to 36 months
  To estimate parameters in the target population associated with molecular testing patterns, including molecular test type
reason for molecular testing | From enrolment to follow-up of up to 36 months
  To estimate parameters in the target population associated with molecular testing patterns, including reason for molecular testing
Molecular testing laboratory type | From enrolment to follow-up of up to 36 months
  To estimate parameters in the target population associated with molecular testing patterns, including molecular testing laboratory type
reason for not performing a molecular test | From enrolment to follow-up of up to 36 months
  To estimate parameters in the target population associated with molecular testing patterns including reason for not performing a molecular test
mutation status | From enrolment to follow-up of up to 36 months
  To estimate parameters in the target population associated with molecular testing patterns including molecular testing result of mutation status
mutation type | From enrolment to follow-up of up to 36 months
  To estimate parameters in the target population associated with molecular testing patterns, including molecular result of mutation type
histologic/phenotypic transformation | From enrolment to follow-up of up to 36 months
  To estimate parameters in the target population associated with molecular testing patterns, including histologic/phenotypic transformation
Overall CNS metastases rate | From enrolment to follow-up of up to 36 months
  Overall CNS metastases rate, defined as the number of patients developing CNS metastases divided by the number of evaluable patients (From start of 2L therapy)
Brain metastases rate | From enrolment to follow-up of up to 36 months
  Brain metastases rate, defined as the number of patients developing brain metastases divided by the number of evaluable patients
Leptomeningeal metastases rate | From enrolment to follow-up of up to 36 months
  Leptomeningeal metastases rate, defined as the number of patients developing leptomeningeal metastases divided by the number of evaluable patients
Type of treatments for CNS metastases | From enrolment to follow-up of up to 36 months
  Treatments for CNS metastases, including type of treatment
Date of treatments for CNS metastases | From enrolment to follow-up of up to 36 months
  Treatments for CNS metastases, including dates of treatment
Change in score from baseline for each QoL domain measured at each subsequent site visit | From enrolment to follow-up of up to 36 months
  To assess patient-reported HRQoL using European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire - Core 30 items (EORTC QLQ-C30) and European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire - Lung Cancer 13 items (EORTC QLQ-LC13)
Change in score from baseline for overall QoL measured at each subsequent site visit | From enrolment to follow-up of up to 36 months
  To assess patient-reported HRQoL using European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire - Core 30 items (EORTC QLQ-C30) and European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire - Lung Cancer 13 items (EORTC QLQ-LC13)

CONTACTS AND LOCATIONS:
Overall Officials: Weimin Li, Doctor, Principal Investigator — West China Hospital
Locations (13):
- China (13):
  - Research Site, Beijing
  - Research Site, Changsha
  - Research Site, Chengdu
  - Research Site, Guangzhou
  - Research Site, Hangzhou
  - Research Site, Harbin
  - Research Site, Hohhot
  - Research Site, Qingdao
  - Research Site, Shenyang
  - Research Site, Suzhou
  - Research Site, Taizhou
  - Research Site, Xi'an
  - Research Site, Zhuji

IPD SHARING:
Plan to Share IPD: No
Chinese laws and regulations do not allow.

REFERENCES:
- [Derived] Tian P, Wu L, Zhou C, Tan J, Wang K, Luo F, Liu Y, Guo Y, Li Y, Liu Z, Gong Y, Wang Y, Xian J, Li W. Molecular testing, treatment patterns, and outcomes in EGFR-mutated non-small cell lung cancer: the PISCES study. Future Oncol. 2025 Aug;21(19):2537-2547. doi: 10.1080/14796694.2025.2529094. Epub 2025 Jul 28. PMID 40717496
- See also: CSR Synopsis_Redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5160R00031&attachmentIdentifier=88ccdb22-f8a3-4496-a2ef-eeeb23bd01fb&fileName=CSR_Synopsis_Redacted.pdf&versionIdentifier=